CLINICAL TRIAL: NCT04972682
Title: Tailoring Postoperative Management Through Sentinel Lymph Node Biopsy in Low- and Intermediate-Risk Endometrial Cancer: a Prospective Open-label Single-arm Clinical Trial
Brief Title: [SENTRY] Tailoring Postoperative Management Through Sentinel Lymph Node Biopsy in Low- and Intermediate-Risk Endometrial Cancer
Acronym: SENTRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow City Oncology Hospital No. 62 (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCOH62-07-08-21
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Endometrial Cancer; Endometrial Neoplasms; Endometrial Adenocarcinoma; Endometrial Cancer Stage I; Endometrial Cancer Stage II; Endometrial Endometrioid Adenocarcinoma; Sentinel Lymph Node; Hysterectomy; Laparoscopic Hysterectomy
Keywords: Endometrial Cancer; Endometrial Adenocarcinoma; Sentinel Lymph Node Biopsy; Laparoscopic Hysterectomy; Adjuvant Therapy; FIGO
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: A single-center prospective open-label single-arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic total hysterectomy with bilateral salpingo-oophorectomy and sentinel lymph node biopsy (Experimental): This arm includes patients with endometrioid adenocarcinoma of the endometrium of low- and intermediate-risk who will undergo a laparoscopic total hysterectomy and bilateral salpingo-oophorectomy with sentinel lymph node biopsy (SLNB) performed with near-infrared-guided surgery using indocyanine green (ICG).
  Interventions: Procedure: Laparoscopic total hysterectomy with bilateral salpingo-oophorectomy and sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Laparoscopic total hysterectomy with bilateral salpingo-oophorectomy and sentinel lymph node biopsy — Laparoscopic total hysterectomy, bilateral salpingo-oophorectomy (BSO), and sentinel lymph node (SLN) biopsy are executed by 1 of 5 experienced gynecologic oncologists. SLN mapping utilizes indocyanine green (ICG) at a standard concentration of 2.5 mg/mL - 1 mL is injected into the cervix at the 3 and 9 o'clock positions (total dose - 5 mg) to a depth of 5-10 mm, initiated right after general anesthesia induction. Diagnostic laparoscopy employs the Image 1S equipment (KARL STORZ©, Tuttlingen, Germany). Upon examination, fluorescence in the near-infrared spectrum is observed. Successful mapping is indicated by identifying a lymphatic vessel with at least one LN. Detected SLNs are then extracted, and the total hysterectomy with BSO is completed. SLN frozen section remains at the surgeon's discretion. If metastasis surfaces in the SLN either during the frozen section or routine assessment, the option for systematic LN dissection in a subsequent procedure exists although not mandatory.

SUMMARY:
While total hysterectomy without lymph node staging is standard for low- and intermediate-risk endometrial cancer, certain histopathologic factors can necessitate additional interventions. Our study assesses the influence of sentinel lymph node (SLN) biopsy on postoperative decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically verified low-grade endometrioid adenocarcinoma of the endometrium (G1-G2)
* FIGO stage IA
* FIGO stage IB and II when LND is contraindicated
* No contraindications for surgery
* Signed informed consent

Exclusion Criteria:

* • Age <18 years
* Presence of tumor spread outside the corpus uteri
* Absence of tumor invasion into the myometrium
* High-grade tumor (G3)
* Bokhman type 2 tumor (e.g., clear cell adenocarcinoma, serous adenocarcinoma, carcinosarcoma, endometrial stromal sarcoma)
* Preoperative treatment of endometrial cancer including radiotherapy, systemic chemotherapy, or hormone therapy
* Prior pelvic or retroperitoneal LND
* History of surgeries on the uterus and uterine appendages, with exceptions such as cesarean section, tubectomy, oophorectomy, ovarian resection, ovarian biopsy, and ovarian cauterization
* Allergy to iodine-containing drugs
* Contraindications to surgical treatment
* Lack of signed informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in postoperative treatment strategy | Up to 3 weeks after surgery
  The rate of change in postoperative treatment based on the SLNB results and postoperative histology (percentage). A change in postoperative treatment strategy is defined as any difference between treatment plans set by the tumor board before and after receiving the SLN biopsy information.

SECONDARY OUTCOMES:
Adjustments in FIGO staging | Up to 3 weeks after surgery
  The rate of change in disease stage based on SLNB results and postoperative histology (percentage).
Bilateral SLN detection | At the end of the surgery - 1 day
  The rate of bilateral SLN detection (percentage).
Details of intraoperative complications of SLN biopsy | At the end of the surgery - 1 day
  The actual list of intraoperative complications associated with SLN mapping and biopsy. They include but are not limited to an intraoperative bleeding, small and large bowel injury, ureter and bladder injury, nerve injury, and allergic reaction to indocyanine green (ICG).
The rate of intraoperative complications of SLN biopsy | At the end of the surgery - 1 day
  Percentage of patients experiencing intraoperative complications associated with SLN mapping and biopsy listed above.
Major postoperative morbidity | Up to 30 days after surgery
  Major postoperative morbidity following the procedure (percentage).
Postoperative mortality | Up to 30 days after surgery
  Postoperative mortality following the procedure (percentage).
Incidence of lymphedema | Up to 24 months after surgery
  The rate of lower extremities lymphedema (percentage).
Pelvic recurrence rate | 24 months after surgery
  The percentage of patients experiencing pelvic recurrence after surgical treatment.
Time to pelvic recurrence | 24 months after surgery
  Time from surgical treatment to detected pelvic recurrence in months.

CONTACTS AND LOCATIONS:
Locations (1):
- 1. Department of Gynecologic Oncology, Moscow City Oncology Hospital No. 62, Istra, Moscow Oblast, Russia

REFERENCES:
- [Result] Sorokin P, Novozhilov M, Utkin D, Abduragimova Z, Dudina I, Nikiforchin A, Kulikova S. Tailoring postoperative management through sentinel lymph node biopsy in low- and intermediate-risk endometrial cancer - the SENTRY clinical trial. Klin Onkol. 2024;38(2):126-133. doi: 10.48095/ccko2024126. PMID 38697821
- See also: The SENTRY clinical trial is a prospective open-label single-arm clinical trial aimed to evaluate the impact of SLN biopsy on the postoperative decision-making process in patients with presumed low- and intermediate-risk endometrial cancer. — https://www.linkos.cz/english-summary/klinicka-onkologie-journal/2024-04-15-2-en/prizpusobeni-pooperacni-lecby-pomoci-biopsie-sentinelove-lymfaticke-uzliny-u-kar-1/